CLINICAL TRIAL: NCT03208166
Title: Pilot Study of Pre-Ischemic Conditioning for Intracranial Atherosclerosis
Acronym: PICASSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of Southern California (Other); University of California, Los Angeles (Other); Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062831
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Ischemic Conditioning (Experimental): Doctormate device is used daily.
  Interventions: Device: Doctormate; Other: Usual Care
- Usual Care (Other): Standard medical care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Doctormate — Ischemic conditioning device
  Arms: Ischemic Conditioning
Other: Usual Care — Standard medical care

SUMMARY:
The purpose of this study is to determine the effects of the Doctormate device, a specialized blood pressure cuff used to perform remote limb ischemic conditioning, on cerebral blood flow in subjects with intracranial atherosclerosis. Previous studies in patients with narrowing of the brain arteries have shown that this device is safe to use and suggested that if this device is inflated in both arms for 5 minutes, followed by deflation for 5 minutes and repeated 4 times in a row every day for 6-9 months, the risk of another stroke is lowered and the device may increase the blood flow to the brain.

DETAILED DESCRIPTION:
In this prospective randomized pilot study, 10 eligible high-risk subjects with ICAS will be randomized to RLIC (bilateral upper extremity daily for 30 days) plus medical management (n=5) or medical management alone (n=5). The medical management, which is the standard of care, will be started at study enrollment and continued until close-out in all subjects. It will consist of aspirin 325 mg per day, clopidogrel 75 mg per day, and risk factor management primarily targeting a systolic BP < 140 mmHg and LDL cholesterol < 70 mg /dl.

All subjects will undergo baseline brain arterial spin labeling (ASL) and perfusion MRI to measure CBF and have blood drawn for biomarkers 3-5 days after randomization to allow for washout of any effect from the test RLIC treatment that will be done prior to randomization to determine the subjects' tolerability to RLIC treatment. The period of 3-5 days will provide flexibility for scheduling these tests. After the baseline MRI and biomarker tests are completed, the subjects randomized to RLIC will begin daily RLIC for 30 days. Each daily RLIC treatment will consist of 4 cycles of 5-minute inflations of both blood pressure cuffs simultaneously to a pressure of 200 mm Hg with 5 minutes of reperfusion between each inflation using the Doctormate device.

All subjects will return for their close-out visits 33-35 days after enrolling in the study and will undergo brain ASL and perfusion MRI and have blood drawn for biomarkers at that visit. The study will be conducted at 4 sites (MUSC, MCG, UCLA, USC) to enable us to evaluate the consistency of CBF measurements across multiple sites and to ensure that the recruitment target of 10 subjects will be met in time to allow for the subsequent NIH grant submission in 2017.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic cerebral infarction within 30 days of enrollment attributed to 70-99% stenosis of a major intracranial artery (carotid artery, MCA stem (M1), vertebral artery, or basilar artery) that is documented by any of the following: MRA, CTA, or catheter angiography. Percent stenosis will be measured according to WASID criteria (= 1 - [Ds / Dn]) x 100% with Ds [diameter of stenosis] and Dn [diameter of normal vessel]).19
2. Modified Rankin score of ≤ 3
3. Age ≥ 30 years and ≤ 90 years. Subjects 30-49 years are required to meet at least one additional criteria (i-vi) provided in the table below to qualify for the study. This additional requirement is to increase the likelihood that the symptomatic intracranial stenosis in subjects 30-49 years is atherosclerotic.

   * i. insulin dependent diabetes for at least 15 years
   * ii. at least 2 of the following atherosclerotic risk factors: hypertension (BP > 140/90 or on antihypertensive therapy); dyslipidemia (LDL > 130 mg /dl or HDL < 40 mg/dl or fasting triglycerides > 150 mg/dl or on lipid lowering therapy); smoking; non-insulin dependent diabetes or insulin dependent diabetes of less than 15 years duration; family history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, peripheral vascular surgery in parent or sibling who was < 55 years of age for men or < 65 for women at the time of the event
   * iii. history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease
   * iv. any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by non-invasive vascular imaging or catheter angiography and is considered atherosclerotic
   * v. aortic arch atheroma documented by non-invasive vascular imaging or catheter angiography
   * vi. any aortic aneurysm documented by non-invasive vascular imaging or catheter angiography that is considered atherosclerotic
4. Recent (within 30 days) negative pregnancy test in a female who has had any menses in the last 12 months
5. Subject is willing and able to return in 30 days for close-out visit for the study
6. Subject is available by phone
7. Subject is able to apply the conditioning device or has access to another person (family member, friend) who can assist with application of conditioning device if needed
8. Subject understands the purpose and requirements of the study, can make him/herself understood, and has provided informed consent
9. Subject is able to undergo brain MRI

Exclusion Criteria:

1. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform one of these procedures
2. Plan to perform concomitant angioplasty or stenting of an extracranial vessel tandem to an intracranial stenosis
3. Intracranial tumor (except meningioma) or any intracranial vascular malformation
4. Thrombolytic therapy within 24 hours prior to enrollment
5. Progressive neurological signs within 24 hours prior to enrollment
6. Any intracranial hemorrhage (parenchmal, subarachnoid, subdural, epidural) within 90 days
7. Any untreated chronic subdural hematoma
8. Intracranial arterial stenosis due to arterial dissection, Moya Moya disease; any known vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with CSF pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; post-partum angiopathy; suspected vasospastic process, suspected recanalized embolus
9. Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction less than 30%
10. History of upper extremity ischemia, known subclavian or brachial artery stenosis, subclavian steal syndrome, any upper extremity soft tissue, orthopedic or vascular injury, or mastectomy or other procedure that may contraindicate taking blood pressure or having a cuff on the arm for the conditioning treatment
11. Difference in systolic blood pressure of > 15 mm Hg between both arms
12. Known allergy to aspirin or clopidogrel
13. Active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets < 100,000, hematocrit < 30, INR > 1.5, clotting factor abnormality that increases the risk of bleeding, current alcohol or substance abuse, uncontrolled severe hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 115 mm Hg), severe liver impairment (AST or ALT > 3 x normal, cirrhosis), subject on dialysis
14. Major surgery (including open femoral, aortic, or carotid surgery, cardiac) within previous 30 days or planned in the next 30 days after enrollment
15. Indication for warfarin or heparin beyond enrollment (NOTE: exceptions allowed for subcutaneous heparin for deep vein thrombosis (DVT) prophylaxis while hospitalized)
16. Diabetic subjects taking sulfonylurea drugs
17. Severe neurological deficit that renders the subject incapable of living independently
18. Dementia or psychiatric problem that prevents the subject from following the protocol reliably
19. Co-morbid conditions that may limit survival to less than 3 months
20. Pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study
21. Claustrophobia requiring sedation for MRI
22. Enrollment in another study that would conflict with the current study

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc I Chimowitz, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ischemic Conditioning | Usual Care
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ischemic Conditioning | Usual Care | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (0) | 46 (0) | 55 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Cerebral Blood Flow (CBF)
Description: Percent change CBF from baseline to 30 days as determined by ASL MRI imaging.
Time Frame: Baseline and 30 days
Measure: Number; unit: percentage increase in CBF
Arm/Group | Ischemic Conditioning | Usual Care
Number analyzed (Participants) | 1 | 1
percentage increase in CBF | 0 | 25

2. Primary Outcome: Change in Putative Blood Biomarkers
Description: Change in the absolute levels of the following biomarkers will be measured from baseline to 30 days: Nitrite, IL-10, SDF1, Micro RNA 144. Lp-PLA2, IL-6. hsCRP, Soluble E selectin, ICAm, MMP-9, PAI-1,tPA, ADMA
Time Frame: 30 days
Population: Since recruitment in the trial was terminated early and there were only 2 patients enrolled, one in the conditioning arm and one in the standard of care arm, a decision was made not to do these experimental biomarkers (which are done in batch) since interpretating the results would be challenging with just one patient in each arm.
Arm/Group | Ischemic Conditioning | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days (the duration of the study)
Arm/Group | Ischemic Conditioning | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Study was stopped early because of low recruitment rate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT03208166/Prot_SAP_000.pdf